CLINICAL TRIAL: NCT03716726
Title: Understanding and Addressing the Social Determinants of Health for Families of Children With Sickle Cell Anemia Within Pediatric Hematology
Brief Title: Sickle Cell Anemia WE CARE
Acronym: SCAWECARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: H-38214; 1R01HL141774-01A1 (NIH)
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Social Determinants of Health; Unmet Social Needs; WE CARE
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Pragmatic pilot cluster RCT to examine the implementation of WE CARE as standard of care in two of the four outpatient pediatric hematology clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-WE CARE (Experimental): The WE CARE SDoH Screening Survey will be given at all visits by the front desk staff to all parents of Sickle Cell Anemia patients who present to the pediatric hematology clinic. They will also be provided the Family Resource Book.
  Clinical team members (i.e. medical assistants and providers) will be trained to review the WE CARE Social Determinants of Health survey at visits and to provide community resource information sheets to parents with needs. The completed surveys will be scanned into the electronic health record (EHR).
  Interventions: Behavioral: WE CARE SDoH Screening Survey; Behavioral: Family Resource Book
- Control-Standard of Care (Experimental): Standard of care for pediatric patients with sickle cell anemia will be delivered.
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: WE CARE SDoH Screening Survey — The survey will be given at all visits by the front desk staff to all parents of SCA patients. It consists of 12 questions designed to: (1) briefly identify 6 unmet material needs (e.g., childcare, employment, food security, household heat, housing inadequate education) by self-report and (2) using a family-centered approach, determine whether parents would like assistance with each problem Parents wanting help will receive a resource referral. Clinical team members will be trained to review the WE CARE SDoH survey at visits and to provide community resource information sheets to parents with needs. Completed surveys will be scanned into the EHR
  Arms: Intervention-WE CARE
Behavioral: Family Resource Book — The Family Resource book will contain one-page information sheets listing community resources (e.g., food pantries) and their contact information (i.e. telephone number) for each specific material need (e.g., food insecurity). Information sheets will be specific to each site and written at, or below, the 8th grade level. For parents with an identified need, providers will be instructed to give an information sheet. The book will contain six separate tabs, one for each unmet need, and will contain multiple copies of the information sheets. The Family Resource Book will be made available in each exam room. The investigators will work with each practice to create a Family Resource Book prior to study initiation.
  Arms: Intervention-WE CARE
Other: Standard of care — Usual outpatient care for pediatric patients with sickle cell anemia will be provided.
  Arms: Control-Standard of Care

SUMMARY:
This mixed-methods study aims to understand the implementation of a previously tested, efficacious social determinants of health (SDoH) screening and referral intervention in the outpatient pediatric hematology setting; qualitatively assess possible mechanisms for such interventions on improving child health; and obtain population-specific empirical estimates to plan a large-scale clinical trial.

DETAILED DESCRIPTION:
Social determinants of health (SDoH)-the conditions in which people are born, grow, work, live, and age-are key drivers of health and health disparities. Children with medical complexity are particularly at-risk given their high healthcare need and utilization. Although the American Academy of Pediatrics and payers such as the Centers for Medicaid and Medicare Services are now recommending medical providers screen for SDoH at visits, studies have not yet demonstrated the impact of SDoH screening and referral interventions on improving child health and have fallen short of exploring potential mechanisms by which such interventions could improve health outcomes. Children with sickle cell anemia (SCA) are an ideal population in which to study the impact of SDoH interventions given the high prevalence of poverty and unmet material needs among this population and the disease's significant morbidity and mortality. This proposal addresses a timely clinically- and policy-relevant research gap by: (1) implementing a SDoH intervention in two outpatient pediatric hematology clinics and gathering preliminary data to assess its impact on child health; and (2) characterizing the potential mechanisms by which addressing SDoH may lead to improved health outcomes. The research team has developed, tested, and implemented a SDOH intervention (WE CARE) which relies on existing clinical processes to screen for unmet material needs and refer parents to community services; efficacy data demonstrates its positive impact on parental receipt of community resources. The investigators now propose conducting a pragmatic pilot cluster randomized controlled trial (RCT) to examine the implementation of WE CARE as standard of care in two of the four hematology clinics. To preliminarily examine outcomes,100 parents of children with SCA (25 per site) will be recruited and followed for one year in order to explore how addressing unmet social needs within the delivery of medical care may improve healthcare utilization and health outcomes. Given the limitations of applying existing theoretical frameworks to culturally diverse populations such as those with SCA, the investigators will also employ a mixed methods approach to characterizing how SDoH influences disease management processes. The specific aims are to: (1) Implement WE CARE in two pediatric hematology clinics in order to field test key study logistics and understand the facilitators and barriers to implementation and accelerate its adoption; (2) Obtain population-specific empirical estimates of study parameters to plan a large-scale multi-site cluster RCT of WE CARE that will definitely assess its impact on improving health outcomes for children with SCA; and (3) Qualitatively assess possible mechanisms linking SDoH interventions to improved health outcomes. It has significant implications for child health policy and is a critical step in potentially transforming the delivery of healthcare for medically complex children.

ELIGIBILITY:
Inclusion Criteria:

* Adult parents of children with SCA (0-12 years of age) who take a daily medication (penicillin or hydroxyurea)to
* English or Spanish speaking

Exclusion Criteria:

* Foster parents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arvin Garg, MD MPH, Principal Investigator — University of Massachusetts Medical School, Worcester
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinics
Groups:
- Intervention-WE CARE: The WE CARE SDoH Screening Survey will be given at all visits by the front desk staff to all parents of Sickle Cell Anemia patients who present to the pediatric hematology clinic. They will also be provided the Family Resource Book.
  Clinical team members (i.e. medical assistants and providers) will be trained to review the WE CARE Social Determinants of Health survey at visits and to provide community resource information sheets to parents with needs. The completed surveys will be scanned into the electronic health record.
  Family Resource Book: The Family Resource book will contain one-page information sheets listing community resources (e.g., food pantries) and their contact information (i.e. telephone number) for each specific material need (e.g., food insecurity). Information sheets will be specific to each site and written at, or below, the 8th grade level. For parents with an identified need, providers will be instructed to give an information sheet. The book will contain six separate tabs, one for each unmet need, and will contain multiple copies of the information sheets. The Family Resource Book will be made available in each exam room.
Period: Completed Baseline Assessment
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Started | 51; 2 Clinics | 61; 2 Clinics
Completed | 41; 2 Clinics | 49; 2 Clinics
Not Completed | 10; 0 Clinics | 12; 0 Clinics
Not completed — Did not complete baseline assessment | 10 | 12
Period: 12 Months Followup
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Started | 41; 2 Clinics | 49; 2 Clinics
Completed | 31; 2 Clinics | 32; 2 Clinics
Not Completed | 10; 0 Clinics | 17; 0 Clinics
Not completed — Lost to Follow-up | 10 | 17

BASELINE CHARACTERISTICS:
Population: Parents of children with sickle cell anemia ages 0-12 years of age taking at least one daily medication who completed baseline assessment.
Groups:
- Intervention-WE CARE: Received WE CARE screener and referral program
- Control-Standard of Care: Received standard of care
- Total: Total of all reporting groups
Arm/Group | Intervention-WE CARE | Control-Standard of Care | Total
Number analyzed (Participants) | 41 | 49 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [33 to 42] | 36 [31 to 39] | 37 [32 to 40]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 29 | 43 | 72
  Male | 7 | 6 | 13
  Unknown | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 30 | 40 | 70
  Unknown or Not Reported | 6 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 36 | 65
  White | 2 | 1 | 3
  More than one race | 2 | 8 | 10
  Unknown or Not Reported | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 41 | 49 | 90
Brief Coping Orientation to Problems Experienced (COPE) Inventory at Baseline [Median (Inter-Quartile Range); unit: scores on a scale] — Self-reported measure of effective and ineffective ways to cope with a stressful life event. 28 total items (list of coping behaviors) scored on a 4-point Likert scale from 1 (I haven't been doing this at all) to 4 (I've been doing this a lot). There are 14 coping behaviors for the 28 items and scores for each of the 14 can range from 1-8.
  scores on a scale
    Self distraction | 3 [2 to 5] | 4 [2 to 5] | 3.5 [2 to 5]
    Active coping | 5 [3 to 6] | 5 [4 to 8] | 5 [3 to 7]
    Denial | 2 [2 to 3] | 2 [2 to 4] | 2 [2 to 3]
    Substance use | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
    Use of emotional support | 4 [2 to 6] | 4 [2 to 5] | 4 [2 to 5]
    Use of instrumental support | 4 [3 to 5] | 4 [2 to 5] | 4 [2 to 5]
    Behavioral disengagement | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
    Venting | 2 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
    Positive reframing | 5.5 [4 to 7] | 5 [2 to 8] | 5 [3 to 7]
    Planning | 4 [3 to 6] | 4 [2 to 6] | 4 [3 to 6]
    Humor | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
    Acceptance | 5.5 [4 to 7] | 5 [4 to 7] | 5 [4 to 7]
    Religion | 6 [3 to 8] | 6 [4 to 8] | 6 [4 to 8]
    Self blame | 2 [2 to 3] | 2 [2 to 4] | 2 [2 to 4]
Patient Health Questionnaire 8 (PHQ-8) [Count of Participants; unit: Participants] — Patient Health Questionnaire depression scale (PHQ-8) is an 8 item instrument with possible responses for each item of 0=Not at all, 1=Several days 2= More than half the days, 3=Nearly every day. The range of scores is 0 to 24, A score of 10 or greater is considered major depression, 20 or more is severe major depression. Population: Parents of children with sickle cell anemia ages 0-12 years of age taking at least one daily medication who completed baseline assessment. Missing PHQ-8 data from 3 participants in WE CARE group.
  Participants
    None (0-9 points): number analyzed (Participants) | 38 | 49 | 87
    None (0-9 points) | 33 | 42 | 75
    Major (10-19 points): number analyzed (Participants) | 38 | 49 | 87
    Major (10-19 points) | 5 | 5 | 10
    Severe (≥ 20 points): number analyzed (Participants) | 38 | 49 | 87
    Severe (≥ 20 points) | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Emergency Department (ED)/Acute Care Visits
Description: Data on number of ED visits and acute care visits abstracted from the EHR.
Time Frame: 12 months
Population: EHR data abstraction was done at 12 months for all participants who completed the baseline assessment.
Measure: Median (Full Range); unit: number of visits
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Number analyzed (Participants) | 41 | 49
number of visits | 0 [0 to 4] | 1 [1 to 10]

2. Primary Outcome: Parental Enrollment in Community Resources
Description: Self-reported enrollment in a new community resource, where "yes" indicates enrollment in a new resource, and "no" indicates no enrollment in a new resource.
Time Frame: 12 months
Population: Data are missing for 3 participants in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Number analyzed (Participants) | 31 | 29
Participants
  Any new resource | 9 | 11
  Child care | 1 | 2
  Employment | 1 | 0
  Housing | 1 | 1
  Food | 1 | 1
  Education | 1 | 2
  Utilities | 5 | 7

3. Secondary Outcome: Personal Health Questionnaire Depression Scale (PHQ-8)
Description: Patient Health Questionnaire depression scale (PHQ-8) is an 8 item instrument with possible responses for each item of 0=Not at all, 1=Several days 2= More than half the days, 3=Nearly every day. The range of scores is 0 to 24. A score of 10 or greater is considered major depression, 20 or more is severe major depression.
Time Frame: 12 months
Population: Data are missing for 1 intervention participant and 4 control participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Number analyzed (Participants) | 30 | 28
Participants
  None (0-9 points) | 28 | 25
  Major (10-19 points) | 1 | 3
  Severe (≥ 20 points) | 1 | 0

4. Secondary Outcome: Brief COPE (Coping Orientation to Problems Experienced Inventory) at 12 Months
Description: Self-reported measure of effective and ineffective ways to cope with a stressful life event. 28 total items (list of coping behaviors) scored on a 4-point Likert scale from 1 (I haven't been doing this at all) to 4 (I've been doing this a lot). There are 14 coping behaviors for the 28 items and scores for each of the 14 can range from 1-8.
Time Frame: 12 months
Population: Data are missing for 1 participant in the intervention arm and 4 participants in the control arm
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Number analyzed (Participants) | 30 | 28
score on a scale
  Self-distraction | 2 [2 to 4] | 3.5 [2 to 5]
  Active copying | 4 [3 to 6] | 5 [2.5 to 6.5]
  Denial | 2 [2 to 2] | 2 [2 to 2.5]
  Substance use | 2 [2 to 2] | 2 [2 to 2]
  Use of emotional support | 3 [2 to 5] | 4 [2 to 6]
  Use of instrumental support | 2 [2 to 2] | 4 [2 to 5]
  Behavioral engagement | 2 [2 to 2] | 2 [2 to 2]
  Venting | 2 [2 to 3] | 2 [2 to 4]
  Positive reframing | 4.5 [2 to 5] | 4 [2.5 to 5]
  Planning | 4 [2 to 6] | 4 [2.5 to 6]
  Humor | 2 [2 to 2] | 2 [2 to 2]
  Acceptance | 6 [3 to 8] | 6 [3.5 to 8]
  Religion | 4.5 [3 to 7] | 6.5 [2.5 to 7.5]
  Self-blame | 2 [2 to 3] | 2 [2 to 3]

5. Secondary Outcome: Vaso-occlusive Episodes
Description: Number of painful vaso-occlusive episodes (VOE) requiring an ED or acute care clinic visit
Time Frame: 12 months
Population: EHR data abstraction was done at 12 months for all participants who completed the baseline assessment.
Measure: Median (Inter-Quartile Range); unit: number of episodes
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Number analyzed (Participants) | 41 | 49
number of episodes | 1 [0 to 1] | 1 [0 to 1]

6. Secondary Outcome: Prescriptions for Sickle Cell Disease
Description: Data on prescriptions written and filled for hydroxyurea and penicillin will be collected through EHR review. . Number of days covered by prescriptions will be reported
Time Frame: 12 months
Population: EHR data abstraction was done at 12 months for all participants who completed the baseline assessment except for 1 participant in the intervention group and for 2 participants in the control group; for those 3 participants the data are missing.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Number analyzed (Participants) | 40 | 47
days
  Penicillin | 365 [30 to 365] | 196 [126 to 331]
  Hydroxurea | 365 [90 to 365] | 258 [126 to 313]

7. Secondary Outcome: Hemoglobin Values Related to Medication Adherence
Description: Laboratory markers commonly affected by hydroxyurea medication from the CBC (complete blood count) include hemoglobin and hemoglobin F levels, white blood cell and absolute neutrophil counts, and mean corpuscular volume. Each wil be abstracted from the medical records.
Time Frame: 12 months
Population: EHR data abstraction was done at 12 months for all participants who completed the baseline assessment.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Number analyzed (Participants) | 41 | 49
g/dL | 9.3 [8.8 to 10] | 8.8 [7.9 to 9.9]

8. Secondary Outcome: White Blood Cell and Absolute Neutrophil Counts Related to Medication Adherence
Description: Laboratory markers commonly affected by hydroxyurea medication from the CBC (complete blood count) including hemoglobin and hemoglobin F levels, white blood cell and absolute neutrophil counts, and mean corpuscular volume. Each will be abstracted from medical records.
Time Frame: 12 months
Population: EHR data abstraction was done at 12 months for all participants who completed the baseline assessment.
Measure: Median (Inter-Quartile Range); unit: cells per dL
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Number analyzed (Participants) | 41 | 49
cells per dL
  White blood cell count (per dL) | 8.6 [6.8 to 12.6] | 9.0 [6.8 to 13.5]
  Absolute neutrophil count (per dL) | 3.5 [2.0 to 5.3] | 3.4 [2.5 to 5.4]

9. Secondary Outcome: Mean Corpuscular Volume Values Related to Medication Adherence
Description: Laboratory markers commonly affected by hydroxyurea medication from the CBC (complete blood count) including hemoglobin and hemoglobin F levels, white blood cell and absolute neutrophil counts, and mean corpuscular volume (MCV) will be abstracted from medical records. MCV is a measure of the average volume of a red blood corpuscle (or red blood cell).
Time Frame: 12 months
Population: EHR data abstraction was done at 12 months for all participants who completed the baseline assessment.
Measure: Median (Inter-Quartile Range); unit: femtoliters (10^15; fl)
Arm/Group | Intervention-WE CARE | Control-Standard of Care
Number analyzed (Participants) | 41 | 49
femtoliters (10^15; fl) | 96 [89.5 to 102.5] | 90.1 [82.6 to 94.9]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention-WE CARE | Control-Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/49
Other Adverse Events (participants affected / at risk) | 0/41 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03716726/Prot_SAP_001.pdf
  • Informed Consent Form (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03716726/ICF_000.pdf